CLINICAL TRIAL: NCT06335784
Title: Mental Imagery and Targeted Memory Reactivation in Insomnia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Lampros Perogamvros, Attending Physician, University Hospital, Geneva
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-00456
Record Dates: First submitted 2024-03-21; First posted 2024-03-28 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Insomnia Disorder
Keywords: Insomnia; Odors; Imagery; TMR
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Odorants

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Sleep Hygiene (SH) (Active Comparator): Participants will receive 4 weekly individual sessions of standardized instructions on sleep hygiene, that they will be asked to apply every day for 4 weeks. Each session will consist of providing patients with advice to help their sleep without any CBT-I or other complementary medicine components. They will also have an odorless diffuser being diffused at the end of each weekly individual session and during the night.
  Interventions: Behavioral: Sleep Hygiene; Other: "Rocking bed" if patients still have insomnia complaints (ISI >10) after the 4 weeks of the intervention
- Imagery Rescripting (IR) (Experimental): Participants will receive 4 weekly individual sessions of IR. The IR technique consists of imagining a negative memory or image as vividly as possible, and of transforming it into a positive one. An odorless diffuser will be presented while imagining the positive imagery generated during IR. During 4 weeks, patients of this group will practice IR at home, every day in bed and have the same odorless diffuser being diffused during the night.
  Interventions: Behavioral: Imagery Rescripting (IR); Other: "Rocking bed" if patients still have insomnia complaints (ISI >10) after the 4 weeks of the intervention
- Targeted Memory Reactivation (TMR) (Experimental): Participants will receive 4 weekly individual sessions of IR, at the end of which, a chosen odor will be presented while imagining the positive imagery generated during IR. During 4 weeks, patients of this group will practice IR at home every day in bed and have the same odor being diffused during the night.
  Interventions: Behavioral: Imagery Rescripting (IR) and Targeted Memory Reactivation (TMR) during sleep; Other: "Rocking bed" if patients still have insomnia complaints (ISI >10) after the 4 weeks of the intervention
- Odor Alone (OA) (Active Comparator): Participants will have a chosen odor diffused during the night for 4 weeks and will receive 4 weekly individual sessions of standardized instructions on sleep hygiene, that they will be asked to apply every day for 4 weeks. The chosen odor will be diffused at the end of each weekly individual session.
  Interventions: Behavioral: Sleep Hygiene + Odor; Other: "Rocking bed" if patients still have insomnia complaints (ISI >10) after the 4 weeks of the intervention

INTERVENTIONS:
Behavioral: Imagery Rescripting (IR) — Imagery rescripting (IR) is a technique where the individual is instructed to imagine a negative memory or image as vividly as possible, and to change it in a direction that he/she desires. IR seems particularly efficient because it is based on the experienced emotions during perceptual information processing, thereby eliciting stronger emotional responses than verbal processing.
  Arms: Imagery Rescripting (IR)
Behavioral: Imagery Rescripting (IR) and Targeted Memory Reactivation (TMR) during sleep — Targeted Memory Reactivation (TMR) is a technique used to strengthen a memory trace during sleep. TMR is used to modify memory formation through the application of cues during sleep. In this TMR protocol, an olfactory cue is associated with the imagery rescripting (IR) during the day, and then administered during sleep. In that way, the replay of the associated memory and its corresponding neural representation in memory networks are artificially promoted, a procedure which usually strengthens memory consolidation. Previous studies have shown that TMR in sleep reduces emotional arousal, making it a promising technique for insomnia.
  Arms: Targeted Memory Reactivation (TMR)
Behavioral: Sleep Hygiene — Sleep hygiene education includes modifications in the behavior (e.g., exercise, coffee, alcohol intake) and environment (e.g., light, noise, temperature conditions) that offer to the individual the foundation for healthy sleep. Sleep hygiene is an important component in treating ID, but insufficient and less effective than CBT-I when offered alone.
  Arms: Sleep Hygiene (SH)
Behavioral: Sleep Hygiene + Odor — Sleep hygiene instructions will be applied in the presence of an odor, which will be also used during the night.
  Arms: Odor Alone (OA)
Other: "Rocking bed" if patients still have insomnia complaints (ISI >10) after the 4 weeks of the intervention — Rocking stimulation boosts brain oscillations in deep sleep (i.e., sleep spindles and slow oscillations) into a rhythmic appearance supporting a neurophysiological mechanism whereby continuous rocking entrains endogenous thalamo-cortical sleep oscillations. The beneficial effects of rocking strengthening the continuity of sleep might have clinical applications and it will be of interest to evaluate if such non-pharmacological could improve sleep and reduce such features of hyperarousal in ID patients.

SUMMARY:
In this clinical trial, the investigators test whether mental Imagery Rescripting (IR), a technique where the individual is instructed to transform a negative memory or image into a positive one, and olfactory Targeted Memory Reactivation (TMR), a technique used to strengthen memories, can reduce hyperarousal and insomnia severity in patients with Insomnia Disorder (ID).

Patients with ID will be randomized into four groups: in the first group (SH group), patients will have 4 weekly sessions (1 session/week) of a minimal intervention for insomnia (sleep hygiene information) in the presence of an odorless diffuser, which will be also used during the night. In the second group (IR group), patients will use IR during wakefulness to induce a state of relaxation and positive emotionality. More specifically, during 4 weekly sessions of IR, patients will imagine a negative scenario related to their pre-sleep images or current concerns (e.g., social interactions, self-image, sleep problem, nightmares) and transform it into a positive script. They will then perform IR every day for 4 weeks at home in the presence of an odorless diffuser, which will be also used during the night. In the third group, patients will undergo the same 4 weekly IR sessions and an odor will be paired to the positive imagery and will be diffused during the night (TMR group). Patients from this group will also perform IR every day for 4 weeks at home. Finally, the fourth group (OA group) will receive 4 weekly sessions of sleep hygiene instructions in the presence of an odor, which will be also used during the night.

Clinical evaluation of insomnia severity before and after the intervention will take place using the Insomnia Severity Index (ISI, primary outcome measure).

At the end of these interventions, patients with persistent symptoms will benefit from an alternative experimental treatment ("rocking bed") in which they will be cradled for one night.

The investigators hypothesize that patients treated with IR will have significantly reduced insomnia severity compared to participants who received a minimal intervention. They also hypothesize that patients of the TMR group, will have more reduced ID severity compared to participants performing IR and with an odorless diffuser, therefore without an association (IR group). Finally, they hypothesize that one night of sleeping in a rocking bed will improve objective measures of sleep in ID compared to a stationary condition.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45 years
* Insomnia disorder according to the International Classification of Diseases 3 (ICSD-3)
* ISI > 10
* PSQI > 5
* No other current treatment for Insomnia

Exclusion Criteria:

* patients with another psychiatric disorder requiring acute treatment according to DSM-5
* patients with medical (e.g. neurological disorders) or other disorders explaining the predominant complaint of insomnia (e.g., sleep apneas with ODI>15/h, restless legs syndrome, periodic limb movements with PLM>15, chronic pain)
* patients with significant substance use/withdrawal
* patients with heavy smoking
* known pregnancy
* patients suffering from anosmia, olfactory related issues and respiratory pathology

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline, 5 Weeks and 3 Months
  Standardized questionnaire that measures ID severity, the score ranges from 0-28, zero indicating no symptom severity and 28 indicating the higher symptom severity.

SECONDARY OUTCOMES:
Pittsburgh sleep quality index (PSQI) | Baseline, 5 Weeks and 3 Months
  Validated self-report scale to assess the quality of sleep, the score ranges from 0-21, zero indicating no symptom severity and 21 indicating the higher symptom severity.
Total Sleep Time (TST) | Baseline and 5 Weeks
  Time from sleep onset to sleep offset. This outcome is measured both subjectively and objectively.
Wake After Sleep Onset (WASO) | Baseline and 5 Weeks
  Number of awakenings during the night. This outcome is measured both subjectively and objectively.
Beck Depression Inventory II (BDI-II) | Baseline, 5 Weeks and 3 Months
  Validated self-report scale to assess depressive symptoms, the score ranges from 0-63, zero indicating no symptom severity and 63 indicating the higher symptom severity.
State Trait Anxiety Inventory (STAI) | Baseline, 5 Weeks and 3 Months
  Validated self-report scale to assess anxiety, the score ranges from 20-80, 20 indicating no symptom severity and 80 indicating the higher symptom severity.
Sleep efficiency (SE) | Baseline and 5 Weeks
  Ratio between total time spent in bed and total sleep time. This outcome is measured both subjectively and objectively.
Micro-arousals | Baseline and 5 Weeks
  Objective measure of micro-awakenings during the night.

OTHER OUTCOMES:
Temperament and Character Inventory | Baseline and 5 Weeks
  A 240-item self-administered questionnaire designed to measure 4 temperament and 3 character scales.
Pre-sleep Arousal Scale (PSAS) | Baseline and 5 Weeks
  A 16-item self-reported questionnaire designed to measure pre-sleep arousability, the score ranges from 16-80, 16 indicating no symptom severity and 80 indicating the higher symptom severity.
Arousal Predisposition Scale (APS) | Baseline and 5 Weeks
  A 12-item self-reported questionnaire designed to measure arousability
Digit Span Task | Baseline and 5 Weeks
  A working memory task, asking the participant to repeat a string of numbers which are displayed verbally, exactly as given, for "digits forward," and in reverse order for "digits backward"
Psychomotor Vigilance Task (PVT) | Baseline and 5 Weeks
  A sustained-attention, reaction-timed task that measures the speed with which subjects respond to a visual stimulus.
Declarative word paired-associate learning task | Baseline and 5 Weeks
  Subjects will be instructed to learn 46 word-pairs with an immediate (pre-sleep) and a delayed one (post-sleep) to assess overnight improvement
Attachment Style Questionnaire (ASQ) | Baseline and 5 Weeks
  A 40-item self-reported questionnaire designed to measure attachment style.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Sleep Medicine, Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No